CLINICAL TRIAL: NCT02012894
Title: Physiopathologic Evaluation of Esophageal Function After Laparoscopic Sleeve Gastrectomy
Brief Title: Laparoscopic Sleeve Gastrectomy and Gastroesophageal Acid Reflux
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Fabrizio Rebecchi, MD, University of Turin, Italy
Other Study IDs: RGEOB/76
Record Dates: First submitted 2013-12-05; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Gastroesophageal Reflux; Obesity
Keywords: Obesity; Gastroesophageal reflux; sleeve gastrectomy; pH-monitoring; manometry
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese patients with preoperative GER: Obese patients selected for laparoscopic sleeve gastrectomy with preoperative GER at 24 H pH-monitoring (Group A)
- Obese patients without preoperative GER: Obese patients selected for laparoscopic sleeve gastrectomy without preoperative GER at 24 H pH-monitoring (Group B)

SUMMARY:
Symptomatic Gastroesophageal Reflux (GER) is considered by many a contraindication to laparoscopic sleeve gastrectomy (LSG). However, of the few studies that have investigated the relationship between LSG and GER the majority reported only changes in symptoms and manometric data, while assessment of GER using 24-hour pH monitoring is lacking.

The aim of this study is to evaluate the effect of LSG on GER in morbidly obese patients.

DETAILED DESCRIPTION:
Consecutive morbidly obese patients selected for LSG are included in a prospective clinical study. Gastroesophageal function is evaluated using a clinical validated questionnaire, upper endoscopy, esophageal manometry and 24-h pH monitoring before and 24 months after LSG.

ELIGIBILITY:
Inclusion Criteria:

* history of obesity exceeding 5 years
* documented previous weight loss attempts,
* body mass index (BMI)) of 40-50 kg/m2
* age of 18-60 years.

Exclusion Criteria:

* contraindications to pneumoperitoneum
* large esophageal hiatal hernia
* pregnancy,
* drug or alcohol abuse,
* psychological disorders (e.g., bulimia, depression)
* hormonal or genetic obesity-related disease,
* previous gastric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive morbidly obese patients selected for LSG
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in DeMeester's score | baseline, 24 months after LSG
  Use of the composite score that evaluates GER at 24-h pH monitoring before and 24 months after LSG. It includes numbers of reflux episodes, upright time in reflux, recumbent time in reflux, total time in reflux, reflux episodes over 5 minutes, longest reflux episodes

SECONDARY OUTCOMES:
Change from baseline in lower esophageal sphincter pressure | baseline, 24 months after LSG
  Esophageal manometry measures several parameters including lower esophageal sphincter pressure
Change from baseline in amplitude of esophageal peristaltic waves | baseline, 24 months after LSG
  Esophageal manometry evaluates quality and amplitude of esophageal peristalsis
Change from baseline in grade of esophagitis | baseline, 24 months after LSG
  Upper endoscopy is performed to assess preoperative and postoperative presence and severity of esophagitis
Change from baseline in Gastroesophageal reflux disease Symptom Assessment Scale score | Baseline, 24 months after LSG
  Standard and validated questionnaire is used to assess gastroesophageal symptoms and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Rebecchi, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- University of Turin, Turin, Turin, Italy

REFERENCES:
- [Background] Tai CM, Huang CK, Lee YC, Chang CY, Lee CT, Lin JT. Increase in gastroesophageal reflux disease symptoms and erosive esophagitis 1 year after laparoscopic sleeve gastrectomy among obese adults. Surg Endosc. 2013 Apr;27(4):1260-6. doi: 10.1007/s00464-012-2593-9. Epub 2012 Dec 12. PMID 23232995
- [Background] Petersen WV, Meile T, Kuper MA, Zdichavsky M, Konigsrainer A, Schneider JH. Functional importance of laparoscopic sleeve gastrectomy for the lower esophageal sphincter in patients with morbid obesity. Obes Surg. 2012 Mar;22(3):360-6. doi: 10.1007/s11695-011-0536-5. PMID 22065341
- [Background] Mahawar KK, Jennings N, Balupuri S, Small PK. Sleeve gastrectomy and gastro-oesophageal reflux disease: a complex relationship. Obes Surg. 2013 Jul;23(7):987-91. doi: 10.1007/s11695-013-0899-x. PMID 23460263
- [Derived] Rebecchi F, Allaix ME, Giaccone C, Ugliono E, Scozzari G, Morino M. Gastroesophageal reflux disease and laparoscopic sleeve gastrectomy: a physiopathologic evaluation. Ann Surg. 2014 Nov;260(5):909-14; discussion 914-5. doi: 10.1097/SLA.0000000000000967. PMID 25379861